CLINICAL TRIAL: NCT01022905
Title: Prospective Cohort Study of the Influence of Age, Underlying Disease and Immunosuppression on Vaccine Responses to Influenza A H1N1/09 Immunization in High-risk Patients.
Brief Title: Vaccine Responses to Influenza A H1N1/09 Immunization in High-risk Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Prof. Claire-Anne Siegrist, University Hospital, Geneva
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CER-09-234
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2010-03-01 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infection; Rheumatic Disease; Cancer; Transplant; Pediatrics
Keywords: HIV infection; transplant; rheumatic disease; cancer; children
MeSH Terms: conditions — HIV Infections; Rheumatic Diseases; Neoplasms | interventions — Vaccines; pandemrix; halofantrine; focetria; lactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-risk patients ( 5 cohorts) (Experimental)
  Interventions: Biological: Adjuvanted influenza A(H1N1) vaccines
- Healthy controls (Active Comparator)
  Interventions: Biological: Adjuvanted influenza A(H1N1) vaccines

INTERVENTIONS:
Biological: Adjuvanted influenza A(H1N1) vaccines — Immunization (1-2 doses)
  Other Names: Pandemrix (GSK); Focetria (Novartis)

SUMMARY:
The objective of this study is to assess vaccine responses to novel adjuvanted influenza A(H1N1) vaccines in patients at high risks of influenza A(H1N1) complications.

DETAILED DESCRIPTION:
This prospective, open-label, parallel-cohorts study will include up to 1250 patients and 250 controls to whom influenza A(H1N1) immunization was recommended.

Six cohort have been established, enrolling patients with HIV infection, rheumatic diseases, organ transplant, cancer, pediatric patients and healthy controls.

Subjects will be assessed for specific antibody responses (all), T cell responses (subset) and solicited vaccine adverse events. Vaccine safety evaluation will include the influence of immunization on underlying diseases (HIV infected patients, patients with auto-immune diseases) or graft function (transplant patients) - as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* medically recommended influenza A(H1N1) immunization
* signed informed consent

Exclusion Criteria:

* failure or refusal to provide sufficient blood for antibody determination

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1141 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Antibody responses (inhibition of hemagglutination) | 4-6 weeks after immunization

SECONDARY OUTCOMES:
Antibody responses (neutralization) | 4-6 weeks after immunization
Vaccine safety : - Solicited adverse events - graft function before / after immunization - influence of immunization on underlying disease (HIV infection, autoimmune diseases) | 4-6 weeks after immunization
T cell responses | 4-6 wks after immunization

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Siegrist CA, van Delden C, Bel M, Combescure C, Delhumeau C, Cavassini M, Clerc O, Meier S, Hadaya K, Soccal PM, Yerly S, Kaiser L, Hirschel B, Calmy A; H1N1 Study Group; Swiss HIV Cohort Study (SHCS). Higher memory responses in HIV-infected and kidney transplanted patients than in healthy subjects following priming with the pandemic vaccine. PLoS One. 2012;7(7):e40428. doi: 10.1371/journal.pone.0040428. Epub 2012 Jul 27. PMID 22848378
- [Derived] Schappi MG, Meier S, Bel M, Siegrist CA, Posfay-Barbe KM; H1N1 Study Group. Protective antibody responses to influenza A/H1N1/09 vaccination in children with celiac disease. J Pediatr Gastroenterol Nutr. 2012 Jun;54(6):817-9. doi: 10.1097/MPG.0b013e318248e7be. PMID 22228003
- [Derived] Mohty B, Bel M, Vukicevic M, Nagy M, Levrat E, Meier S, Grillet S, Combescure C, Kaiser L, Chalandon Y, Passweg J, Siegrist CA, Roosnek E; Blood and Marrow Transplant Program; Geneva University Hospitals H1N1 study group. Graft-versus-host disease is the major determinant of humoral responses to the AS03-adjuvanted influenza A/09/H1N1 vaccine in allogeneic hematopoietic stem cell transplant recipients. Haematologica. 2011 Jun;96(6):896-904. doi: 10.3324/haematol.2011.040386. Epub 2011 Mar 21. PMID 21422117
- [Derived] Meier S, Bel M, L'huillier A, Crisinel PA, Combescure C, Kaiser L, Grillet S, Posfay-Barbe K, Siegrist CA; H1N1 Epidemiology Study Group of Geneva. Antibody responses to natural influenza A/H1N1/09 disease or following immunization with adjuvanted vaccines, in immunocompetent and immunocompromised children. Vaccine. 2011 Apr 27;29(19):3548-57. doi: 10.1016/j.vaccine.2011.02.094. Epub 2011 Mar 17. PMID 21419775
- [Derived] Gabay C, Bel M, Combescure C, Ribi C, Meier S, Posfay-Barbe K, Grillet S, Seebach JD, Kaiser L, Wunderli W, Guerne PA, Siegrist CA; H1N1 Study Group. Impact of synthetic and biologic disease-modifying antirheumatic drugs on antibody responses to the AS03-adjuvanted pandemic influenza vaccine: a prospective, open-label, parallel-cohort, single-center study. Arthritis Rheum. 2011 Jun;63(6):1486-96. doi: 10.1002/art.30325. PMID 21384334